CLINICAL TRIAL: NCT00010361
Title: Study of Total Body Irradiation and Fludarabine Followed By Allogeneic Peripheral Blood Stem Cell or Bone Marrow Transplantation in Combination With Cyclosporine and Mycophenolate Mofetil in Patients With Inherited Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15577; FHCRC-1475.00; NCT00144742 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-02 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2006-08

CONDITIONS: Metabolism, Inborn Errors; Granulomatous Disease, Chronic
MeSH Terms: conditions — Metabolism, Inborn Errors; Granulomatous Disease, Chronic | interventions — Cyclosporine; fludarabine; Mycophenolic Acid

INTERVENTIONS:
Drug: cyclosporine
Drug: fludarabine
Drug: mycophenolate mofetil

SUMMARY:
OBJECTIVES: I. Determine the safety of total body irradiation and fludarabine followed by allogeneic peripheral blood stem cell or bone marrow transplantation in combination with cyclosporine and mycophenolate mofetil for establishing mixed chimerism in patients with inherited disorders.

II. Determine whether this regimen can establish mixed chimerism in these patients.

III. Determine whether mixed chimerism is sufficient to reverse disease symptoms in these patients.

IV. Determine the safety of donor lymphocyte infusions to eliminate persistent disease in these patients with mixed chimerism.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive fludarabine IV over 2 hours on days -4 to -2 followed by total body irradiation and peripheral blood stem cell or bone marrow transplantation on day 0. Patients also receive oral or IV cyclosporine 2-3 times daily on days -3 to 50 (related donor) or 100 (unrelated donor) and oral mycophenolate mofetil twice daily on days 0 to 28 (related donor) or 40 (unrelated donor).

Patients may also receive donor lymphocyte infusion for continued treatment of symptoms in the event of mixed chimerism and in the absence of graft-versus-host disease.

Patients are followed weekly for 1 month, monthly for 2 years, and then annually thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Inherited disorders treatable with allogeneic peripheral blood or bone marrow transplantation At high risk for regimen related toxicity with a conventional transplant
* No severe CNS involvement of disease, defined by IQ score less than 70
* HLA matched donor Sibling donors must be a confirmed match at HLA-A, B, and DRB1 Other related and non-related donors must be matched at HLA-A, B, C, DRB1, and DQB1 A donor homozygous for one allele only at HLA-A, B, C, DRB1, or DQB1 allowed (1 antigen mismatch for graft-versus-host disease, 0 antigen mismatch for graft-rejection)

--Prior/Concurrent Therapy--

* No concurrent growth factors with mycophenolate mofetil

--Patient Characteristics--

* Age: Under 55
* Performance status: Not specified
* Life expectancy: At least 100 days
* Hematopoietic: Not specified
* Hepatic: No evidence of synthetic dysfunction No severe cirrhosis
* Renal: Not specified
* Cardiovascular: LVEF at least 30% No poorly controlled hypertension on multiple antihypertensives
* Other: No organ dysfunction that would preclude survival Not pregnant or nursing Fertile patients must use effective contraception during and for 12 months following study

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2000-11; Primary Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Woolfrey, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States